CLINICAL TRIAL: NCT02012556
Title: A Phase 1 Study to Evaluate the Pharmacokinetics and the Pharmacodynamics of TH9507 Administered Subcutaneously Once Daily for 14 Consecutive Days in HIV Positive Patients
Brief Title: Pharmacokinetic and Pharmacodynamic Study of TH9507, a Growth Hormone-Releasing Factor Analog, in HIV Positive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theratechnologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH9507-CTR-1015
Record Dates: First submitted 2013-11-26; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: HIV
MeSH Terms: interventions — tesamorelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tesamorelin (Experimental)
  Interventions: Drug: Tesamorelin

INTERVENTIONS:
Drug: Tesamorelin
  Other Names: Egrifta

SUMMARY:
The primary objective of the study is to determine the PK (tesamorelin) and PD (IGF-1) profiles of tesamorelin after a single 2 mg subcutaneous administration and after repeated administration once daily for 14 consecutive days. Secondary objectives include the evaluation of the safety and tolerability of tesamorelin following multiple subcutaneous injections.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female, smoker or non-smoker, ≥18 and ≤65 years of age.
* HIV-positive with CD4 cell counts >100 cells/mm3 and viral load <10 000 copies/mL.
* On stable antiretroviral therapy (ART) regimen for at least 8 weeks prior to the first study drug administration.
* Body mass index (BMI) ≥ 20.0 kg/m2.

Main Exclusion Criteria:

* Opportunistic infection or HIV-related disease within 3 months prior to study drug administration.
* History of malignancy of any organ or tissue (with the exception of basal cell carcinoma of the skin, in situ carcinoma of the cervix and stable Kaposi not having required treatment for the past 6 months).
* For male subjects, suspicion of prostate cancer.
* For female subjects, history of breast cancer or strong family history (first degree relative) of breast cancer.
* Known hypopituitarism, history of pituitary tumor/surgery, head irradiation or severe head trauma that had affected the somatotropic axis.
* Use of any experimental or marketed GH or GRF/GHRH products, GH secretagogues, IGF-1, or insulin-like growth factor binding protein-3 (IGFBP-3) within 6 months prior to study drug administration and throughout the study.
* Positive pregnancy test at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Area under the Plasma Concentration versus Time Curve (AUC) of Tesamorelin. | Pre-dose on Days 1, 7, 12, 13, and 14, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, and 4 hours post-dose on Day 1, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, 4, 12, and 24 hours post-dose on Day 14.
Peak Plasma Concentration (Cmax) of Tesamorelin. | Pre-dose on Days 1, 7, 12, 13, and 14, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, and 4 hours post-dose on Day 1, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, 4, 12, and 24 hours post-dose on Day 14.
Time to Maximum Plasma Concentration (Tmax) of Tesamorelin. | Pre-dose on Days 1, 7, 12, 13, and 14, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, and 4 hours post-dose on Day 1, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, 4, 12, and 24 hours post-dose on Day 14.
Apparent Elimination Half-life (T1/2 el) of Tesamorelin. | Pre-dose on Days 1, 7, 12, 13, and 14, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, and 4 hours post-dose on Day 1, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, 4, 12, and 24 hours post-dose on Day 14.
Plasma Clearance (CI/F) of Tesamorelin. | Pre-dose on Days 1, 7, 12, 13, and 14, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, and 4 hours post-dose on Day 1, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, 4, 12, and 24 hours post-dose on Day 14.
Apparent Volume of Distribution (Vd/F) of Tesamorelin. | Pre-dose on Days 1, 7, 12, 13, and 14, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, and 4 hours post-dose on Day 1, and at 0.05, 0.1, 0.15, 0.2, 0.25, 0.333, 0.5, 0.667, 1, 1.33, 2.5, 4, 12, and 24 hours post-dose on Day 14.
Insulin-like Growth Factor-1 (IGF-1) Level at Day 1. | Day 1.
Insulin-like Growth Factor-1 (IGF-1) Level at Day 7 | Day 7.
Insulin-like Growth Factor-1 (IGF-1) Level at Day 13. | Day 13.
Insulin-like Growth Factor-1 (IGF-1) Level at Day 14. | Day 14.

SECONDARY OUTCOMES:
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm Montreal, Montreal, Quebec, Canada